CLINICAL TRIAL: NCT02762682
Title: A Study of Vitamin B12 Status in Children With Infantile Tremor Syndrome and Pre Infantile Tremor Syndrome
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Chaudhary Himanshi, Junior resident, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: Its12pgi
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Infant Nutrition Disorder
MeSH Terms: conditions — Infant Nutrition Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CASES OF ITS AND PRE ITS: 1. Either sex, age less than 3 years
  2. Clinical diagnosis of Infantile Tremor Syndrome as evidenced by the following features:
  [Developmental delay or regression WITH history of exclusive or predominant breast feeding WITH two or more of the following; skin pigmentation, hair depigmentation, tremors] ITS:1 and 2 plus tremors PreITS:1 and 2 without tremors
- HEALTHY CONTROLS: Developmentally normal child not suffering from any acute or chronic neurological illness

SUMMARY:
PRIMARY OBJECTIVES

• To describe the vitamin B12 status in children with infantile tremor syndrome(ITS) and Pre ITS

SECONDARY OBJECTIVES

* To study the vitamin B12 status in mothers of children with infantile tremor syndrome (ITS) and Pre ITS
* To study the blood levels of folate in children with infantile tremor syndrome (includes Pre ITS) and their mothers.

DETAILED DESCRIPTION:
Materials and methods

STUDY SETTING: Hospital based study (Advanced Pediatrics Centre, PGIMER) STUDY PERIOD: July 2015 to December 2016 STUDY DESIGN: Cross sectional, Observational Enrolment criteria Inclusion criteria (cases)

1. Either sex, age less than 3 years
2. Clinical diagnosis of Infantile Tremor Syndrome as evidenced by the following features:

[Developmental delay or regression WITH history of exclusive or predominant breast feeding WITH two or more of the following; skin pigmentation, hair depigmentation, tremors] ITS:1 and 2 plus tremors PreITS:1 and 2 without tremors Exclusion criteria (cases)

1. Parents refusing consent
2. Later confirmation of an alternative diagnosis
3. Patient has received oral or injectable Vitamin B12 in the past 6 months Controls (C)- Normally developing children

   * Inclusion criteria Developmentally normal child not suffering from any acute or chronic neurological illness
   * Exclusion criteria

1.Parent/individual refusing consent 2.Patient has received oral or injectable Vitamin B12 in the past 6 months

PLAN OF THE STUDY All consecutive patients who present in Pediatric Emergency and OPD in Advanced pediatric Centre with suspected Infantile tremor syndrome will be screened for inclusion in the study. Those found eligible would be included after an informed consent. Baseline clinical and demographic profile will be recorded on a proforma..The study aims at assessment of vitamin B12 status in children with ITS. The various manifestations of the syndrome, the presentations, the clinical picture, the development profile, various haematological and biochemical markers would be studied in a detailed manner and recorded on a proforma (annexure).

The first section of the proforma is targeted at the clinical picture of the disease. The presenting features will be recorded. The presenting complaints which can be anything ranging from an episode of upper respiratory tract infection to an apparently healthy child presenting with delayed milestones. A brief history of the development milestones achieved under gross motor, fine motor, language and social milestones is important and form a basis for screening the developmentally delayed children .A feeding history will be taken and is important as this disease is more frequently seen in children who are exclusively/predominantly breastfed. A detailed examination of the child would be done and the findings recorded. Skin and hair changes are very classical of this disease and hence will be to be studied and recorded in detail. A neurological examination will be done to study the neurological status of the children and presence of any extrapyramidal symptoms. Hematological indices will be recorded. Plasma Vitamin B 12, folate, homocysteine levels will be studied.Urine methylmalonic acid along with TMS/GCMS will also be done as a part of this project. Other investigations will be done as per case profile. Any other investigation if done for the case as a part of the treatment or diagnostic evaluation like liver function tests, renal function tests , EEG, CT, MRI will also be recorded.

The second section of the proforma consists of assessment of health and nutritional status of the mother. It aims at establishing any direct relation between the maternal health and development of ITS like picture in their children. Mother's dietary history will be taken to find out whether the maternal diet is lacking in Vitamin B12 and folate. A targeted neurological examination will be done to look for neurological manifestations of vitamin B12 deficiency in form of posterior column tract sensation and presence of peripheral neuropathy. A lab estimation of maternal Vitamin B12,folate and homocysteine levels will also be done and recorded.

Blood samples: Sampling would be done along with routine sampling as far as possible to avoid additional pricks to the child. Plasma would be immediately separated and stored and tested for Vitamin B12 ,homocysteine, methylmalonic acid and folate levels. This blood would be taken from sample already taken for other tests to be done in the child. Confidentiality of records would be maintained. The study is purely observational and will not influence the management of the child. Though as a standard policy all children with ITS would receive Vitamin B12, folate and other supplements and diet counseling will be done.

Blood TMS-acylcarnitine and propionylcarnitine along with evaluation of urine methyl malonic acid as a part of GCMS will also be studied in cases and controls.

Mother's blood samples will also be taken after explaining to them the entire aims and objectives of the study and taking full free voluntary informed consent from them. This would also benefit the mothers in a way because those identified with a deficiency will be given supplements to overcome the deficiency.

Control samples will be taken from children of the same age group admitted for some other ailment. A 2 ml sample will be taken from sample already drawn for other tests to be done in the child. The controls also stand to be benefitted because all children found deficient will be advised Vitamin B12 and folate supplementation immediately.

Vitamin B12 and folate levels will also be studied in the mothers of the 50 controls. All mothers found deficient will be advised Vitamin B12 and folate.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria (cases)

  1. Either sex, age less than 3 years
  2. Clinical diagnosis of Infantile Tremor Syndrome as evidenced by the following features:

     [Developmental delay or regression WITH history of exclusive or predominant breast feeding WITH two or more of the following; skin pigmentation, hair depigmentation, tremors] ITS:1 and 2 plus tremors PreITS:1 and 2 without tremors

     Controls (C)- Normally developing children

     • Inclusion criteria Developmentally normal child not suffering from any acute or chronic neurological illness

     Exclusion Criteria:

     Exclusion criteria (cases)

  <!-- -->

  1. Parents refusing consent
  2. Later confirmation of an alternative diagnosis
  3. Patient has received oral or injectable Vitamin B12 in the past 6 months
* • Exclusion criteria(controls)

  1. Parent/individual refusing consent
  2. Patient has received oral or injectable Vitamin B12 in the past 6 months

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Hospital based study (Advanced Pediatrics Centre, PGIMER) all cases of infantile tremor syndrome (ITS) and pre ITS presenting to APC during the study period
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
vitamin b12 status in children with ITS and preITS | July 2015 to December 2016
  The blood levels of vitamin B-12 and folate would be expressed as mean ± 2 SD or median (range) and will be compared between the children (with infantile tremor syndrome) and their mothers with controls.

SECONDARY OUTCOMES:
vitamin B12 Status in mothers of children with ITS and preITS folate status in these children and their mothers | July 2015 to December 2016
  The blood levels of folate would be expressed as mean ± 2 SD or median (range) and will be compared between the children (with infantile tremor syndrome) and their mothers with controls

CONTACTS AND LOCATIONS:
Overall Officials: Dr Naveen Sankhyan, MBBS,MD,DM, Study Director — PGIMER Chandigarh
Locations (1):
- PGIMER, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chaudhary H, Verma S, Bhatia P, Vaidya PC, Singhi P, Sankhyan N. Infantile Tremor Syndrome or a Neurocutaneous Infantile B12 Deficiency (NIB) Syndrome? Indian J Pediatr. 2020 Mar;87(3):179-184. doi: 10.1007/s12098-019-03117-w. Epub 2020 Jan 27. PMID 31984470